CLINICAL TRIAL: NCT05181956
Title: Testing and Epidemiology of Delta Hepatitis Among Asian Americans
Brief Title: Testing and Epidemiology of Delta Hepatitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asian Pacific Liver Center at Coalition of Inclusive Medicine (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IN-US-980-6356
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Chronic Hepatitis D Infection With Hepatitis B

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study is to

1. Understand the pattern of hepatitis delta screening among medical providers for Asian patients with chronic hepatitis B
2. Determine the proportion of Asian hepatitis B patients who have been screened and who have chronic hepatitis delta
3. Determine the pattern of hepatitis delta screening after education of medical providers on hepatitis delta

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) affects more than 257 million people world-wide with two-thirds of CHB infected people living in Asia and Sub-Saharan Africa. Although the overall prevalence of CHB is high in Asia, the regional prevalence varies; ranging from less than 0.5% in Japan to greater than 12% in Vietnam and Cambodia. Hepatitis delta virus (HDV) is a satellite virus that can infect individuals with hepatitis B virus (HBV) infection to the extent that at least 15-20 million people are conservatively estimated to be chronically infected with HBV and HDV. Chronic HBV/HDV infection is associated with more rapid progression to cirrhosis and a higher incidence of hepatocellular carcinoma (HCC) compared to patients with CHB mono-infection. Prevalence of chronic HBV/HDV remains high in Mongolia, the Mediterranean and Sub-Saharan countries and in the Amazon basin but the true prevalence remains to be determined among many populations and demic groups. Asian Americans are the fastest-growing minority group in the United States, comprising a heterogeneous population from more than 60 different ethnic groups speaking more than 100 different languages, exhibiting substantial socioeconomic diversity. While Asian Americans account for more than 60% of CHB infection in the United States, CHB prevalence varies among the ethnic groups. Similarly, prevalence of chronic hepatitis C and genotype distribution are different among the various Asian groups, underscoring the importance of disaggregating ethnic populations in hepatitis research. We recently reported the high prevalence of HDV infection among Mongolians living in Southern California. However, HDV infection among other Asian-American groups has not been studied, largely because outside of Mongolia and pockets in Vietnam, chronic HBV/HDV infection in Asia appears to below.

Recommendations for routine screening for HDV from various major professional liver societies are not consistent. Asian Pacific Association for the Study of the Liver (APASL) and the European Association for the Study of the Liver (EASL) recommend HDV screening for all HBsAg positive individuals. The American Association for the Study of Liver Diseases recommend testing of HBsAg positive individuals with "low or undetectable HBV DNA but high ALT levels", "persons who inject drugs, men who have sex with men, and immigrants from areas of high HDV with endemicity". However, the accurate prevalence of HDV infection in Asia is not well characterized.

To address this gap in knowledge, there is an important need to accurately characterize prevalence, clinical testing patterns and the epidemiology of HDV infection among disaggregated Asian-American groups.

This study will be conducted in 3 parts. The first part will involve a survey of hepatitis delta (HDV) testing practices among 100-125 physicians and other health care providers that have high volumes of Asian CHB patients. Special care will be made to include physicians and health care providers for patients across different Asian ethnic communities. Almost 45% of U.S. Asians live in the West with 30% residing in California alone. Chinese, Filipinos, Vietnamese and Koreans account for the 4 largest Southeast Asian groups but there are large communities of Thais, Cambodians and Burmese in Southern California and Hmongs in Central California. With over 150,000 Armenians residing in Los Angeles, this is another ethnic group that will be studied. Asian Pacific Liver Center (APLC) has worked closely with community CHB health care providers in previous studies and will build on these collaborations. In addition, APLC plans to collaborate with physicians from Texas (Vietnamese), Minnesota (Hmong) and New York City (Chinese, Koreans). In addition, physicians and providers from other settings will be surveyed; academic (USC, UCLA, Cedars-Sinai, Loma Linda, UCSD, UCSF, Stanford, NYU, Mount-Sinai, University of Hawaii, Southwestern, University of Minnesota) and large managed care organization (Southern California Kaiser, Veterans Administration and Sutter Health). Response to this survey will provide an overview of current practice of HDV testing and management among health care professionals with high numbers of Asian CHB patients and also develop a collaboration for subsequent objectives. Each survey responder will be asked to participate in the second and third parts of the study. Each responder will be individually engaged by the PI with respect to the association of hepatitis delta and chronic hepatitis B and the current guidelines and standards of practice for HDV testing among all CHB patients.

The second part involves a chart review of 50-60 physicians and other providers who follow a minimum of 100 CHB patients in their practice. A retrospective chart review will be performed of all 18 years and older CHB patients with the collection of demographic and clinical data including HDV testing results. These results will be compared with estimates based on physicians' responses to the survey. The data extraction will be performed by trained research coordinators familiar with chart reviews of CHB patients. The quality of data will be regularly monitored by the PI and Mimi Chang DNP (who has conducted CHB studies for more than 10 years).

The third part of the study involves prospectively testing all HDV-untested CHB patients which is the recommendation of APASL and EAS and therefore the standard of care for Asian CHB patients. Participating HCPs will be educated regarding the current recommendations for hepatitis delta testing in patients with chronic hepatitis B, but they will not be coerced to perform hepatitis delta testing nor will hepatitis delta testing be a requirement for participation in the study.

Since CHB patients should be evaluated at least every 6 months, all 18 years and older CHB patients in this study should be captured during the 12-month period of the study. The combined data from part 2 and 3 will be used to calculate the prevalence of HDV among the disaggregated Asian CHB patients. The demographic and clinical characteristics of HDV-CHB co-infected patients will be compared to CHB mono-infected patients. During this study there will be ample opportunity to educate those providing care on the current guidelines for management of CHB patients, which includes testing for HDV.

The study protocol, documentation, data, and all other information generated will be held in strict confidence. Data will be collected at multiple sites with procedures designed to ensure the data's accuracy, confidentiality, and security. The PI will assign participating healthcare providers a site number. Identifying information for the providers will be accessed and stored at a secure locked location accessible to only APLC study team members and destroyed upon completion of the study. Identifiable data for the CHB patients will not be collected by assigning a unique numeric identifier. In addition, carefully specified procedures will be adhered to in all aspects of data collection, analysis, and management throughout the study. Standardized rules for entering data will be maintained to ensure the uniformity of data. Patients' data will be entered into a central database at APLC, with a secured access code. As APLC receives data from the participating sites, only the authorized study team members will log in and review the records for completeness and data accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older chronic hepatitis B patients

Exclusion Criteria:

* 17 years and younger chronic hepatitis B patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years and older chronic hepatitis B patients
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-03 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence rate of chronic HDV | 12 months
  Measure prevalence rate of chronic HDV among disaggregated Asian CHB patients through retrospective and prospective testing
Characteristics of Asian patients with chronic HDV | 12 months
  Describe demographic and clinical characteristics of Asian patients with chronic HDV

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Pacific Liver Center, Los Angeles, California, United States